CLINICAL TRIAL: NCT03865147
Title: An Open, Randomised, Parallel Group Controlled, Single Centre Safety Study to Assess the Safety and Efficacy of Tri-Solfen in Providing Anaesthesia Prior to Surgical Debridement of Leg Ulcers and Post-operative Pain Relief
Brief Title: Single-centre Study to Investigate Safety and Efficacy of Tri-Solfen in Wound Debridement
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Ethics UK Ltd (Industry)
Collaborators: ProTherax Ltd (Unknown); Welsh Wound Innovation Centre Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TriSolfen_H_01; 2018-000613-21 (EudraCT Number)
Record Dates: First submitted 2018-05-02; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Wounds Injuries; Anesthesia, Local
MeSH Terms: conditions — Wounds and Injuries | interventions — Lidocaine; Bupivacaine; Epinephrine; Cetrimonium; Lidocaine, Prilocaine Drug Combination; Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Phase IIA, open, randomised, single and parallel group, therapy controlled single centre study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1 open, pilot phase (Experimental): A pilot group of 10 patients who will receive Tri-Solfen only (non-randomised) once, prior to debridement
  Interventions: Drug: Tri-Solfen Gel (Lidocaine HCl, Bupivacaine HCl, Adrenaline Acid Tartrate /Cetrimide)
- Phase 2 - Tri-Solfen (Experimental): A group of 20 patients who will receive EMLA cream (60 minute application) to anaesthetise the leg ulcer prior to surgical wound debridement, followed on completion of surgery by a single application of Tri-Solfen.
  Interventions: Drug: Tri-Solfen Gel (Lidocaine HCl, Bupivacaine HCl, Adrenaline Acid Tartrate /Cetrimide); Drug: EMLA cream
- Phase 2 - Standard Care (Active Comparator): A group of 20 patients who will receive EMLA Cream (60 minute application) to anaesthetise the leg ulcer prior to surgical wound debridement, followed on completion of surgery by standard of care post-operative analgesia.
  Interventions: Drug: EMLA cream; Drug: Post Operative Analgesia (Paracetamol, Ibuprofen)
- Phase 3 - Tri-Solfen (Experimental): A group of 20 patients who will receive two applications of Tri-Solfen (2mL/10cm2), once prior to debridement and once on completion of the procedure.
  Interventions: Drug: Tri-Solfen Gel (Lidocaine HCl, Bupivacaine HCl, Adrenaline Acid Tartrate /Cetrimide); Drug: Post Operative Analgesia (Paracetamol, Ibuprofen)
- Phase 3 - EMLA (Active Comparator): A group of 20 patients who will receive EMLA Cream (60-minute application) prior to surgical debridement
  Interventions: Drug: EMLA cream; Drug: Post Operative Analgesia (Paracetamol, Ibuprofen)

INTERVENTIONS:
Drug: Tri-Solfen Gel (Lidocaine HCl, Bupivacaine HCl, Adrenaline Acid Tartrate /Cetrimide) — Investigational Drug
  Arms: Phase 1 open, pilot phase; Phase 2 - Tri-Solfen; Phase 3 - Tri-Solfen
Drug: EMLA cream — Active Comparator
  Arms: Phase 2 - Standard Care; Phase 2 - Tri-Solfen; Phase 3 - EMLA
Drug: Post Operative Analgesia (Paracetamol, Ibuprofen) — Standard of Care
  Arms: Phase 2 - Standard Care; Phase 3 - EMLA; Phase 3 - Tri-Solfen

SUMMARY:
This is a Phase IIa open, randomised, single and parallel group, therapy controlled, single centre study, which has been divided into 3 sequential phases, which are designed to study respectively, (a) the time taken to achieve surface anaesthesia, (b) the extent of post-operative pain relief and (c) the depth and quality of anaesthesia during a leg ulcer surgical debridement procedure

DETAILED DESCRIPTION:
As part of the study, patients with leg ulcers (venous, arterial, mixed aetiology or lymphoedema) requiring surgical debridement will attend 4 visits to the study centre (Day 0, Day 1, Day 7 and Day 14). After informed consent and screening for inclusion / exclusion criteria patients will be managed as follows:

Phase 1 (N=10 patients): This is a pilot (non-comparative) phase designed to assess safety, pharmacokinetics and achievement of clinically acceptable levels of surface analgesia for Tri-Solfen in the intended patient population, prior to surgical wound debridement. Prior to surgical debridement all patients will have a single application of the Tri-Solfen product 2mL/10cm2 wound area) administered. The product will be allowed to remain in contact with the wound bed for 1 minute and surface anaesthesia will then be tested by needle-stick for up to 30 minutes after application (at 1, 3, 5, 10, 20 and 30 minutes, i.e. testing will stop when the needle stick can no longer be felt). In parallel serial blood draws of 10mL will be taken at 2min, 30min, 1 hr, 2hrs and 6hrs after application to determine systemic absorption of lidocaine and bupivacaine.

Surgical debridement will proceed after a needle stick can no longer be felt and will cease when either the wound bed is deemed to be clean and free from necrotic tissue in the presence of punctate bleeding or where pain increases to an unacceptable level as defined by the patient. Pain assessments will be carried out during the procedure and at 2 min, 30 min, 1 hour, 6 hrs and 24 hours after the procedure is complete.

Phase 2 (N=40 patients; 20 per group): This is a comparative phase of Tri-Solfen vs standard of care in the management of post-operative analgesia. All patients will receive standard of care (i.e. 60 mins of EMLA Cream) to anaesthetise the leg ulcer and will undergo surgical debridement after a needle stick can no longer be felt and will cease when either the wound bed is deemed to be clean and free from necrotic tissue in the presence of punctate bleeding or where pain increases to an unacceptable level as defined by the patient.

On completion of surgical debridement, patients will be randomised to one of two groups:

* Group 1: a single application of Tri-Solfen (2mL/10cm2) with standard of care post-surgical analgesia (e.g. paracetamol, NSAID or opiate) provided as required (N=20), or
* Group 2: standard of care post-surgical analgesia (e.g. paracetamol, NSAID or opiate) as required only (N=20).

Serial blood draws of 10mL from the Tri-Solfen group will be taken at 2min, 30min, 1 hr, 2hrs and 6hrs after application of Tri-Solfen to determine systemic absorption of lidocaine and bupivacaine. Pain assessments and extent of analgesia required will also be carried out at 2 min, 30 min, 1 hour, 6 hrs and 24 hours.

Phase 3 (N=40 patients; 20 per group). Since debridement of the wound may result in removal of surface anaesthesia, this phase is intended to compare the quality of anaesthesia from standard of care (single application of EMLA cream from administration over 60 minutes) with one application of Tri-Solfen administered pre-surgical debridement, and one application on completion of surgery. Safety and quality of anaesthesia / analgesia in the intended patient population before, during and after the surgical debridement procedure will be monitored.

Prior to debridement, patients will be randomised to either:

* Group 1: Tri-Solfen (2mL/10cm2) administered once prior to wound debridement and once on completion of surgical debridement (N=20)
* Group 2: EMLA cream (1-2g /10cm2). administered to the wound for 60 minutes under an occlusive dressing (N=20).

In both groups, the time taken to achieve clinically acceptable surface anaesthesia required to perform the surgical procedure will be assessed using a needle-stick at the wound site. In patients receiving Tri-Solfen, this will be performed at 1, 3, 5, 10, 20 and 30 minutes after application of the Tri-Solfen - assessments will stop when the needle can no longer be detected by the patient. Needle stick testing will also be undertaken immediately following removal of EMLA cream after 60 minutes in EMLA-treated patients to provide a baseline comparator of pre-operative anaesthetic efficacy.

Surgical debridement will proceed only after a needle stick can no longer be felt and will cease when either the wound bed is deemed to be clean and free from necrotic tissue in the presence of punctate bleeding or where pain increases to an unacceptable level as defined by the patient. Pain assessments will be carried out during the procedure and at 2 min, 30 min, 1 hour, 6 hrs and 24 hours after the procedure is complete.

Serial blood draws of 10mL from the Tri-Solfen group will be taken at 2min, 30min, 1 hr, 2hrs and 6hrs after application of the first dose of Tri-Solfen to determine systemic absorption of lidocaine and bupivacaine from multiple dosing.

All Phases Patients will be followed up for two weeks to confirm that the use of the Tri-Solfen (or EMLA) product do not adversely affect wound healing and to assess the incidence of adverse events, including wound infections

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged over 18 years of age, with a chronic leg ulcer of arterial, venous, mixed aetiology or lymphoedema willing and able to provide informed consent and comply with study procedures.
* Presence of slough, necrotic or unhealthy tissue that requires removal by surgical (sharp) debridement
* Study wound that is 2-30 cm2 in regards surface area and has been present for 1-60 months.
* Presence of acute, non-cyclic pain experienced by the patient following a previous debridement. A baseline pain score (prior to any administration of treatment) should be >50mm on a 100mm visual analogue scale

Exclusion Criteria:

* Patients with an acute or chronic infectious skin disease
* Wound bed with exposed bone, tendon or fascia
* Patients with any anaesthetic allergy or intolerance of local anaesthetics or hypersensitivity to any of the ingredients of the Tri-Solfen or EMLA product
* Patients with cellulitis and/or osteomyelitis
* Patients with porphyria
* Patients with abnormal thyroid function including thyrotoxicosis
* Patients with established ventricular fibrillation, cardiac dilatation (severe angina pectoris, obstructive cardiomyopathy), coronary insufficiency, including angina, organic brain disease or atherosclerosis.
* Patients with clinically significant hepatic or renal insufficiency (glomerular filtration rate <30mL per minute)
* Patients receiving more than 2 week's treatment with immunosuppressive agents in the past 3 months.
* Patients receiving oral corticosteroid therapy or topical corticosteroid on the leg where the reference ulcer is located.
* Any investigational drug use within 30 days
* Severe malnutrition, as judged by the investigator
* Patients who, in the opinion of the investigator, have an existing condition that would compromise their partcipation and follow up in this study
* Patients who have, or are suspected of having any underlying or skin malignancy, or who have received treatment for any active malignancy, apart from non-melanomatic skin cancer, within 3 months prior to treatment.
* History of radiation at the study site
* Any other conditions that could impede wound healing
* Patients receiving concomitant medicines including, Carbemazepines, Rifampicin, Phenytoin, Griseofulvin, Phenobarbitone, and Sulphonylureas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Lidocaine Maximum Plasma Concentration | Day 0 - Day 1
  Blood draws to determine systemic levels of lidocaine
Bupivacaine Maximum Plasma Concentration | Day 0 - Day 1
  Blood draws to determine systemic levels of bupivacaine
Local tolerability assessments | Day 0 - Day 1
  Numerical Rating Scale (0-4) for itch, burn, pain, oedema, exudate, inflammation
Local tolerability assessments | Day 0 - Day 1
  Numerical Rating Scale (0-1) for presence of bleeding and wound infection

SECONDARY OUTCOMES:
Pain on Application | 1 minute
  Numerical Rating Scale (0-3) of none, mild, moderate, severe
Time taken to achieve clinically acceptable surface anaesthesia | 0-30 minutes after application
  Perception of needle-stick at the wound site
Pain during wound debridement | 10-15 minutes
  Verbal pain assessment by the patient during wound debridement
Clinical adequacy of wound debridement | On completion of surgery
  Percentage of wound debrided
Duration of post-operative pain relief | Up to 24 hours
  Assessment of the duration of post-operative pain relief using a VAS

CONTACTS AND LOCATIONS:
Overall Officials: Keith Harding, Principal Investigator — Welsh Wound Innovation Centre
Locations (1):
- Welsh Wound Innovation Centre, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No